CLINICAL TRIAL: NCT01513304
Title: Chiropractic Manual Therapy in Infantile Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Jennifer Bolton (Other)
Responsible Party: Sponsor-Investigator, Professor Jennifer Bolton, Director of Research, Anglo-European College of Chiropractic
Organization: Anglo-European College of Chiropractic (Other)
Purpose: Treatment
Other Study IDs: AECCRCT1
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chiropractic manual therapy (Experimental)
  Interventions: Procedure: Manual therapy

INTERVENTIONS:
Procedure: Manual therapy

SUMMARY:
Efficacy of chiropractic manual therapy in infants with excessive crying behaviour. Influence of parental bias in reporting crying behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Excessive crying,
* infant less than 8weeks of age,
* born at gestational age 37 weeks or later, otherwise healthy

Exclusion Criteria:

* Not accepted for chiropractic care

Max Age: 8 Weeks | Sex: All
Age Groups: Child
Dates: Start 2007-09; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Daily crying diary

CONTACTS AND LOCATIONS:
Locations (1):
- AECC, Bournemouth, Dorset, United Kingdom